CLINICAL TRIAL: NCT05009316
Title: Impact of Social Support and Coping Strategies on the Development and Evolution of Post-Surgical Pain
Brief Title: Impact of Social Support and Coping Strategies on Post-Surgical Pain
Acronym: POPQUEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: POPQUEST
Record Dates: First submitted 2021-08-16; First posted 2021-08-17 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Social Support; Coping Behavior; Post-Surgical Pain, Chronic
Keywords: Pain, Chronic
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Questionnaires (Experimental): Patients will answer online surveys containing different questionnaires that will evaluate psychosocial variables as well as pain variables.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Online-based questionnaires

SUMMARY:
The purpose of the study is to evaluate the impact of social support and pain coping strategies in the development and evolution of post-surgical pain.

DETAILED DESCRIPTION:
This is a longitudinal study. After giving their informed consent, patients will answer online questionnaires assessing pain and different psychosocial variables at these time points: before surgery, one to three days after surgery, and one, three, and six months after surgery.

The psychosocial variables evaluated are the following ones :

* Depression,
* Anxiety,
* Stress,
* Pain Coping Strategies,
* Social Support,
* Couple Support.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years of age.
* Capacity to understand and voluntarily sign an informed consent form in French.

Exclusion Criteria:

* Insufficient French language skills.
* History of psychotic disease.
* History of neurodegenerative pathology.
* History of neurological disease (e.g. stroke)
* Pre-existing pain condition related to the reason for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Intensity of acute post-surgical pain | Three days after surgery
  Questions from the Short Form of the Brief Pain Inventory (translated in French) will be used to assess the intensity of the pain on a numeric rating scale (from 0 to 10) during the three days following surgery.
Development of Persistent post-surgical pain, 3 months | 3 months after surgery
  Using the Short Form of the Brief Pain Inventory, pain will be assessed at three months to determine whether patients will have developed chronic pain.
Persistent post-surgical pain, 6 months | 6 months after surgery
  Using the Short Form of the Brief Pain Inventory, pain intensity will be assessed at 6 months.
Pain interference | 6 months after surgery
  Using the Short Form of the Brief Pain Inventory, pain interference on daily activities will be assessed at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: André Mouraux, Ph.D, Study Chair — Université Catholique de Louvain
Locations (1):
- Institute of NeuroScience (IONS) - UCLouvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No